CLINICAL TRIAL: NCT06274645
Title: Intravascular Ultrasound Guidance for Complex High-Risk Indicated Procedures China Registry
Brief Title: IVUS CHIP China Registry
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IVUS CHIP China Registry
Record Dates: First submitted 2024-01-12; First posted 2024-02-23 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Complex Higher Risk Indicated Patients Undergoing PCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: The OptiCross High Definition (60 MHz) and OptiCross (40MHz) Intravascular Ultrasound (IVUS) catheter from Boston Scientific — The IVUS-guided PCI procedure includes the use of IVUS before PCI (highly recommended) and after PCI (mandatory)

SUMMARY:
The goal of this observational study is to learn about in patients with complex coronary lesions undergoing PCI. The main question[s] it aims to answer are: the clinical efficacy and safety of an IVUS-guided approach in patients with complex coronary lesions undergoing PCI, as well as clinical outcomes up to 2 years. Participants will be treated with IVUS-guided PCI.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years of age
2. Patients with an indication for PCI of at least one lesion satisfying any of the following criteria:

   1. Angiographic heavy calcification
   2. Ostial lesions
   3. True bifurcation lesions involving side-branches >2.5mm
   4. Left main lesions
   5. Chronic total occlusion
   6. In-stent restenosis
   7. Long-lesions (estimated stent length > 28mm) OR Patient with an indication for PCI for any lesion and in need for elective mechanical circulatory support assisted PCI
3. Presenting with silent ischemia, stable angina, unstable angina or non-ST-elevation acute coronary syndrome (NSTE-ACS)
4. All lesions must be suitable for treatment with 2nd generation drug eluting stents (or drug-coated balloons when indicated, e.g., in-stent restenosis, branching of bifurcation lesions)
5. The patient is willing and able to cooperate with registry procedures and follow-up until registry completion
6. Subject is able to confirm understanding of risks, benefits and treatment alternatives and he/she provides informed consent prior to any protocol-related procedure, as approved by the appropriate Ethics Committee

Exclusion Criteria:

1. ST-elevation myocardial infarction or cardiogenic shock within prior 7 days
2. Known untreated severe valvular heart disease
3. Requiring PCI in a diseased aorto-coronary bypass
4. Known contraindication or hypersensitivity to anticoagulants
5. Absolute contraindications or allergy that cannot be pre-medicated, to iodinated contrast or to antiplatelet drugs, including both aspirin and P2Y12 inhibitors
6. Non-cardiac co-morbidities with a life expectancy less than 1 year
7. Currently participating in a clinical trial that is not yet at its primary endpoint. The patient is not allowed to participate in an investigational device or drug study until the trial primary endpoint time point is achieved and may only be enrolled once in the study
8. Women who are pregnant or who are breastfeeding
9. Subject's circumstances that will not allow appropriate consenting procedures or follow-up activities (per investigator's discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IVUS-guided approach in patients with complex coronary lesions undergoing PCI
Sampling Method: Non-Probability Sample
Enrollment: 2020 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Time-to-first-event analysis of these three event including cardiac death, target vessel myocardial infarction will be primarily used for clinical endpoints. | 1 Year
  Target-vessel failure defined as a composite of cardiac death, target vessel myocardial infarction*, or clinically indicated target-vessel revascularization at 1 year. It means the time of the patient's occurrence of any of the three events in one year.

SECONDARY OUTCOMES:
Time-to-first-event analysis will be primarily used for clinical endpoints. | full-time process until 2 Year
  1. The time of the first event of Composite of target-vessel myocardial infarction* and clinically indicated target vessel revascularization
  2. The time of the first event of Clinically-indicated target vessel revascularization
  3. The time of the first event of Composite of cardiac death and target-vessel myocardial infarction*
  4. The time of the first event of Target-Lesion Failure (TLF) defined as a composite of cardiac death, target vessel myocardial infarction*, or clinically indicated target-lesion revascularization
  5. The time of the first event of Target-lesion revascularization
  6. The time of Cardiac death

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
Currently,All data of projects will be shared with sponsors and leading site principal investigators. Other site investigators are undecided.